CLINICAL TRIAL: NCT04633564
Title: Multicenter, Double-Blind, Randomized, Parallel-Group Study to Assess the Efficacy and Safety of MYL-1402O Compared With Avastin®, in the First-line Treatment of Patients With Stage IV Non-Squamous Non-Small Cell Lung Cancer
Brief Title: MYL-1402O Compared With Avastin®, in Patients With Stage IV nsNSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYL-1402O-3001
Record Dates: First submitted 2020-11-02; First posted 2020-11-18 (Actual); Results first posted 2021-02-01 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Multicenter, Double-Blind, Randomized, Parallel-Group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MYL-1402O (Experimental): Patients will begin Period 1 receiving bevacizumab combination therapy (MYL-1402O15 mg/kg IV + Carboplatin AUC 6 IV+ Paclitaxel 200 or 175 mg/m2 IV) on Day 0 of Cycle 1 for up to 6 cycles of therapy. Each cycle will consist of 3 weeks (21 days ± 3 days) and a cycle will start with the administration of bevacizumab (as MYL-1402O ).
  In Period 2, eligible patients will continue to receive bevacizumab ( MYL- 1402O) every 3 weeks as monotherapy.
  Interventions: Biological: Bevacizumab as MYL-1402O
- Avastin (Active Comparator): Patients will begin Period 1 receiving bevacizumab combination therapy ( Avastin15 mg/kg IV + Carboplatin AUC 6 IV+ Paclitaxel 200 or 175 mg/m2 IV) on Day 0 of Cycle 1 for up to 6 cycles of therapy. Each cycle will consist of 3 weeks (21 days ± 3 days) and a cycle will start with the administration of bevacizumab (as Avastin).
  In Period 2, eligible patients will continue to receive bevacizumab (Avastin) every 3 weeks as monotherapy.
  Interventions: Biological: Bevacizumab as Avastin

INTERVENTIONS:
Biological: Bevacizumab as MYL-1402O — Bevacizumab as MYL-1402O 15 mg/kg IV + Carboplatin AUC 6 IV+ Paclitaxel 200 or 175 mg/m2 IV
  Arms: MYL-1402O
Biological: Bevacizumab as Avastin — Bevacizumab as Avastin 15 mg/kg IV + Carboplatin AUC 6 IV+ Paclitaxel 200 or 175 mg/m2 IV
  Arms: Avastin

SUMMARY:
Assess the Efficacy and Safety of MYL-1402O Compared with Avastin®, in the First-line Treatment of Patients with Stage IV Non-Squamous Non-Small Cell Lung Cancer

DETAILED DESCRIPTION:
MYL-1402O is a monoclonal antibody currently being developed by Mylan GmbH, as a proposed biosimilar to European Union and US licensed Avastin (hereafter referred to as Avastin), which is approved as first line treatment in combination with carboplatin and paclitaxel (CP) for patients with Stage IV unresectable, recurrent or metastatic nsNSCLC. This randomized equivalence study is designed to meet the global regulatory requirement for approval of a biosimilar product. For this study, both MYL-1402O and Avastin are considered investigational medicinal products (IMP).

ELIGIBILITY:
Key Inclusion Criteria:

1. Written and signed informed consent
2. Male or female at least 18 years of age with documented imaging diagnosis of Stage IV unresectable, recurrent or metastatic nsNSCLC with at least one measurable lesion as defined by RECIST 1.1
3. Documented histologic or cytologic diagnosis of advanced nsNSCLC with negative or unknown sensitizing epidermal growth factor receptor (EGFR) mutation, and negative or unknown echinoderm microtubule-associated protein like 4 anaplastic lymphoma kinase (EML4 ALK) rearrangement.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
5. Has not received any prior systemic therapy for first-line treatment of advanced lung cancer, except adjuvant chemotherapy, and remained disease-free for at least 12 months from time of surgery, and at least 6 months from last dose of chemotherapy.
6. Treated and stable brain metastasis.

Key Exclusion Criteria:

1. Documented squamous NSCLC or small cell type or large cell neuroendocrine histology
2. History of significant hemoptysis, central tumors with proximity to large vessels and tumor with cavitation
3. Received prior treatment with paclitaxel, bevacizumab or anthracycline or had known hypersensitivity to any of these components.
4. Recent significant cardiac condition or vascular event or inadequately controlled hypertension.
5. On anticoagulant therapy not considered stable
6. Risk of hemorrhage in the central nervous system
7. Recent history of surgery, nonhealing wound, active ulcer, or untreated bone fracture.
8. History of gastrointestinal fistula, perforation, or abscess.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen A Idris, MD, Study Director
Locations (102):
- Belarus (5):
  - Grodno Clinical Regional Hospital, Grodno, Hrodzenskaya Voblasts
  - Mogilev Regional Oncology Dispensary, Minsk, Minsk Oblast
  - Babruysk Interregional Oncological Dispensary, Babruysk
  - State Institution NN Alexandrov Republican Scientific and Practical Centre of Oncology And Medical R, Minsk
  - Grodno Clinical Regional Hospital, Mogilev
- Bosnia and Herzegovina (4):
  - Clinical Hospital Mostar, Mostar
  - Clinical Center University of Sarajevo, Sarajevo
  - Javna zdravstvena ustanova bolnica Trebinje, Trebinje
  - County Hospital Zenica, Zenica
- Bulgaria (2):
  - Complex Oncology Center-Veliko Tarnovo, Veliko Tarnovo
  - Complex Oncology Center - Vratsa EOOD, Vratsa
- Croatia (3):
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Sibenik, Šibenik
  - Clinical Hospital Center Zagreb - PPDS, Zagreb
- Georgia (2):
  - Research Institute of Clinical Medicine, Tbilisi
  - LTD High Technology Medical Center University Clinic, Tbilisi
- Hungary (5):
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Veszprem Megyei Tudogyogyintezet, Farkasgyepü
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktató Kórház, Miskolc
- India (31):
  - City Cancer Center, Vijayawada, Andhra Pradesh
  - Mahatma Gandhi Medical College and Hospital, Visakhapatnam, Andhra Pradesh
  - Regional Cancer Centre Indira Gandhi Institute of Medical Sciences, Patna, Bihar
  - HCG Cancer Center, Ahmedabad, Gujarat
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - Synexus Affiliate - Apple Hospital, Surat, Gujarat
  - Unique Hospital - Multispeciality & Research Institute, Surat, Gujarat
  - Aadhar Health Institute, Hisar, Haryana
  - BGS Global Hospital, Bangalore, Karnataka
  - Sri Venkateshwara Hospital, Bangalore, Karnataka
  - Shetty's Hospital, Bengaluru, Karnataka
  - Amravati Cancer Foundation Sujan Surgical and Cancer Hospital, Amravati, Maharashtra
  - United CIIGMA Institute of Medical Sciences Pvt.Ltd., Aurangabad, Maharashtra
  - Seth Nandlal Dhoot Hospital, Aurangabad, Maharashtra
  - Government Medical College, Nagpur, Maharashtra
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Acharya Tulsi Regional Cancer Institute and Research Centre, Bikaner, Rajasthan
  - Malpani Multispecialty Hospital, Jaipur, Rajasthan
  - Institute of Respiratory Diseases (Chest and TB Hospital), Jaipur, Rajasthan
  - Apex Hospital, Jaipur, Rajasthan
  - Bhagwan Mahaveer Cancer Hospital and Research Centre, Jaipur, Rajasthan
  - Rajiv Gandhi Government General Hospital, Chennai, Tamil Nadu
  - Meenakshi Mission Hospital and Research Center, Madurai, Tamil Nadu
  - Shatabdi Superspeciality Hospital, Lucknow, Uttar Pradesh
  - Chittaranjan National Cancer Institute, Kolkata, West Bengal
  - KLES Dr Prabhakar Kore Hospital and Medical Research Centre, Belagāve
  - Prince Aly Khan Hospital Mumbai, Mumbai
  - Jaslok Hospital and Research Centre, Mumbai
  - Sahyadri Speciality Hospital, Pune
  - Kailash Cancer Hospital and Research Centre, Vadodara
- Ospedale Felice Lotti De Pontedera, Pontedera, Italy
- Philippines (2):
  - Philippine General Hospital, Manila, National Capital Region
  - Cardinal Santos Medical Center, San Juan City, National Capital Region
- Poland (2):
  - Med-Polonia Sp. z o.o., Poznan
  - Radomskie Centrum Onkologii, Radom
- Romania (7):
  - Medisprof SRL, Cluj-Napoca, Cluj
  - Ploiesti Municipal Hospital, Ploieşti, Prahova
  - Spitalul Judetean de Urgenta Sf. Pantelimon Focsani, Focşani, Vrancea
  - Elias Emergency University Hospital, Bucharest
  - Prof. Dr. Alexandru Trestioreanu Oncologic Institute, Bucharest
  - Spitalul Clinic Judetean de Urgenta Sf. Apostol Andrei Constanta, Constanța
  - Oncology Center Sfantul Nectarie, Craiova
- Russia (20):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk
  - Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk
  - Kaluga Regional Oncology Dispensary, Kaluga
  - Republican Clinical Oncology Dispensary of Ministry of Healthcare of Tatarstan Republic, Kazan'
  - Kursk Regional Oncology Centre, Kursk
  - Vitamed, Moscow
  - City Clinical Hospital #1, Novosibirsk
  - Clinical Oncology Dispensary, Omsk
  - Stavropol Regional Clinical Oncology Centre Pyatigorsk Affiliate, Pyatigorsk
  - Ryazan State Medical University n.a. I.P. Pavlov, Ryazan
  - Research Institute of Phtisio-pneumology, Saint Petersburg
  - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Railway Clinical Hospital JSC RZhD, Saint Petersburg
  - Clinical Theoretical and Practical Center of Specialized Kinds of Medical Care, Saint Petersburg
  - Scientific Research Institute of Oncology n.a. N.N. Petrov, Saint Petersburg
  - City Clinical Oncology Dispensary, Saint Petersburg
  - Mordovia State University, Saransk
  - Research Oncology Institute of Tomsk Scientific Center, Tomsk
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
  - Regional Clinical Oncology Hospital, Yaroslavl
- Spain (2):
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - Hospital Son Llatzer, Palma de Mallorca
- Taiwan (4):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - E-DA hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Mackay Memorial Hospital-Taipei branch, Taipei
- Turkey (Türkiye) (2):
  - Gazi University Medical Faculty Gazi Hospital, Ankara
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
- Ukraine (6):
  - Municipal Institution City Clinical Hospital #4 of Dnipro City Council - PPDS, Dnipropetrovsk
  - Municipal Institution SubCarpathian ClinicalOncological Centre, Ivano-Frankivsk
  - MI Kryvyi Rih Oncology Dispensary of Dnipropetrovsk Regional Council, Kryvyi Rih
  - Municipal non profit enterprise of Sumy Regional Council Sumy Regional Clinical Oncology Dispensary, Sumy
  - MNPE Central City Clinical Hospital of Uzhhorod City Council, Uzhhorod
  - MI of Zaporizhzhia Regional Council Zaporizhzhia Regional Clinical Oncology Dispensary, Zaporizhzhia
- Vietnam (4):
  - Bach Mai Hospital, Hanoi
  - National Cancer Hospital, Hanoi
  - National Lung Hospital, Hanoi
  - Cho Ray Hospital, Ho Chi Minh City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 671 subjects enrolled at 89 sites across Eastern Europe, Russia, Asia Pacific, South East Asia.
  Date of first patient randomized: 21 Jan 2017 Date of last patient randomized: 31 Jan 2019
Pre-assignment Details: A total of 1016 patients were screened; 345 patients were screen failures. Most common reasons for screen failures were; 57=met exclusion criteria tumor location in contact with major vessels, 46= withdrew consent; 37= patients who have brain metastasis which was treated and stable at the time of signing ICF and 36= patients did not have at least 1 measurable lesion as defined by RECIST 1.1.
Groups:
- MYL-1402O: Patients will begin Period 1 receiving bevacizumab combination therapy (MYL-1402O15 mg/kg IV + Carboplatin AUC 6 IV+ Paclitaxel 200 or 175 mg/m2 IV) on Day 0 of Cycle 1 for up to 6 cycles of therapy. Each cycle will consist of 3 weeks (21 days ± 3 days) and a cycle will start with the administration of bevacizumab (as MYL-1402O ).
  In Period 2, eligible patients will continue to receive bevacizumab ( MYL- 1402O) every 3 weeks as monotherapy.
  Bevacizumab as MYL-1402O: Bevacizumab as MYL-1402O 15 mg/kg IV + Carboplatin AUC 6 IV+ Paclitaxel 200 or 175 mg/m2 IV
- Avastin: Patients will begin Period 1 receiving bevacizumab combination therapy ( Avastin15 mg/kg IV + Carboplatin AUC 6 IV+ Paclitaxel 200 or 175 mg/m2 IV) on Day 0 of Cycle 1 for up to 6 cycles of therapy. Each cycle will consist of 3 weeks (21 days ± 3 days) and a cycle will start with the administration of bevacizumab (as Avastin).
  In Period 2, eligible patients will continue to receive bevacizumab (Avastin) every 3 weeks as monotherapy.
  Bevacizumab as Avastin: Bevacizumab as Avastin 15 mg/kg IV + Carboplatin AUC 6 IV+ Paclitaxel 200 or 175 mg/m2 IV
Period: Period 1
Arm/Group | MYL-1402O | Avastin
Started | 335 | 329
Completed | 227 | 220
Not Completed | 108 | 109
Not completed — Adverse Event | 28 | 19
Not completed — Death | 8 | 7
Not completed — Lost to Follow-up | 3 | 5
Not completed — Physician Decision | 4 | 12
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Progressive disease | 47 | 51
Not completed — Terminated by Sponsor | 8 | 6
Period: Period 2
Arm/Group | MYL-1402O | Avastin
Started | 200 | 199
Completed | 107 | 102
Not Completed | 93 | 97
Not completed — Adverse Event | 3 | 4
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 4
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Progressive Disease | 74 | 82
Not completed — Terminated by Sponsor | 9 | 3

BASELINE CHARACTERISTICS:
Population: The primary efficacy endpoint was the ORR as assessed by an independent review during the first 18 Weeks, according to RECIST 1.1. The primary endpoint was analyzed differently to meet the requirements of FDA and EMA. For FDA, the primary efficacy endpoint was based on the ratio of ORRs and for EMA it was based on difference in ORRs.
Groups:
- Total: Total of all reporting groups
Arm/Group | MYL-1402O | Avastin | Total
Number analyzed (Participants) | 337 | 334 | 671
Age, Categorical [Count of Participants; unit: Participants] — Population: 7 patients are Baseline failures (Randomized but Screen failed at Baseline visit) and not dosed.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 237 | 236 | 473
    >=65 years | 100 | 98 | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (9.60) | 59.2 (9.73) | 59.3 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 123 | 247
  Male | 213 | 211 | 424
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 226 | 232 | 458
  Race: Asian | 111 | 102 | 213
Region of Enrollment [Number; unit: participants]
  Romania | 3 | 4 | 7
  Hungary | 15 | 14 | 29
  Philippines | 1 | 1 | 2
  Ukraine | 86 | 74 | 160
  Belarus | 12 | 12 | 24
  India | 99 | 92 | 191
  Russia | 65 | 75 | 140
  Spain | 2 | 1 | 3
  Vietnam | 10 | 7 | 17
  Turkey | 1 | 1 | 2
  Taiwan | 1 | 2 | 3
  Poland | 3 | 2 | 5
  Georgia | 28 | 30 | 58
  Bulgaria | 3 | 4 | 7
  Bosnia and Herzegovina | 8 | 11 | 19
  Croatia | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Analysis of Overall Response Rate ( ORR) of MYL-1402O as Compared to Avastin
Description: The primary efficacy endpoint Overall Response Rate (ORR) will be based on best tumor responses as assessed by an independent review at any time point during the first 18 weeks, and assessed according to RECIST 1.1. The primary efficacy analysis is based on the ratio of the MYL-1402O ORR to the Avastin ORR at Week 18 based on the Intent to Treat ( ITT) set of patients.
Time Frame: 18 weeks after first dosing per patient
Population: The primary efficacy analysis was conducted in the Intent To Treat population (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | MYL-1402O | Avastin
Number analyzed (Participants) | 337 | 334
Participants
  Responders | 140 | 144
  Non-Responders | 197 | 190
Statistical Analysis 1: Comparison: MYL-1402O vs Avastin; Test type: Equivalence — The equivalence region is (0.73, 1.36); Risk Ratio (RR) = 0.96, 90% CI 2-sided [0.83 to 1.12]

ADVERSE EVENTS:
Time Frame: Active collection period of AEs will be from the time the patient signs the ICF through the Safety Follow Up Visit. Pre-existing diseases or conditions (reported at time of screening) will not be considered AEs unless there is an increase in the frequency or severity, or a change in the quality of the disease or condition. Progression of NSCLC and its consequences will not be collected as an AE even if they lead to hospitalization or meet any other seriousness criteria including death.
Description: The Investigator is responsible for the detection and documentation of events meeting the criteria and definition of an AE or SAE. At each visit, the patient will be allowed time to spontaneously report any issues since the last visit or evaluation. The Investigator will then monitor and/or ask about or evaluate AEs using non-leading questions. Any clinically relevant observations made during the visit are also to be considered AEs.
Arm/Group | MYL-1402O | Avastin
All-Cause Mortality (participants affected / at risk) | 101/335 | 82/329
Serious Adverse Events (participants affected / at risk) | 59/335 | 55/329
Other Adverse Events (participants affected / at risk) | 311/335 | 304/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MYL-1402O (N=335) | Avastin (N=329)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 7 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 6
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Sepsis (Infections and infestations) | 3 | 2
Pneumonia (Infections and infestations) | 3 | 1
Gastroenteritis (Infections and infestations) | 3 | 0
Infectious Pleural Effusion (Infections and infestations) | 2 | 1
Peritonitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 0 | 1
Eye Infection Fungal (Infections and infestations) | 0 | 1
Gastroenteritis Salmonella (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 0 | 1
Rectal Abscess (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric Perforation (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Peptic Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cardicac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure Acute (Cardiac disorders) | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
COR Pulmonale Acute (Cardiac disorders) | 1 | 0
Coronary Artery disease (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Ventricular Arrhythmia (Cardiac disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Venous Thrombosis (Vascular disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Impaired Healing (General disorders) | 0 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1
Cererovascular accident (Nervous system disorders) | 2 | 1
Cerebral Small Vessel Ischamic Disease (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 | 1
Pyelocalieectasis (Renal and urinary disorders) | 0 | 1
Renal Cyst Ruptured (Renal and urinary disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Angle Closure Glaucoma (Eye disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MYL-1402O (N=335) | Avastin (N=329)
Anaemia (Blood and lymphatic system disorders) | 111 | 112
Thrombocytopenia (Blood and lymphatic system disorders) | 104 | 80
Neutropenia (Blood and lymphatic system disorders) | 68 | 76
Leukopenia (Blood and lymphatic system disorders) | 38 | 41
Alopecia (Skin and subcutaneous tissue disorders) | 148 | 168
Peripheral Sensory Neuropathy (Nervous system disorders) | 74 | 66
Headache (Nervous system disorders) | 26 | 17
Hypoaesthesia (Nervous system disorders) | 15 | 20
Nausea (Gastrointestinal disorders) | 56 | 49
Vomiting (Gastrointestinal disorders) | 54 | 38
Diarrhoea (Gastrointestinal disorders) | 46 | 30
Stomatitis (Gastrointestinal disorders) | 22 | 8
Asthenia (General disorders) | 53 | 33
Pyrexia (General disorders) | 31 | 21
Fatigue (General disorders) | 26 | 27
Alanine Aminotranferase Increased (Investigations) | 25 | 29
Aspartate Aminotransferase Increased (Investigations) | 22 | 19
Weight decreased (Investigations) | 22 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 23
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 18
Decreased Appetite (Metabolism and nutrition disorders) | 43 | 32
Hypertension (Vascular disorders) | 19 | 16
Proteinuria (Renal and urinary disorders) | 11 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT04633564/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT04633564/SAP_001.pdf